CLINICAL TRIAL: NCT06983184
Title: Menstrual Cycle-Synced Neuromuscular Training
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sophia Ulman (Other)
Collaborators: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor-Investigator, Sophia Ulman, PhD, Texas Scottish Rite Hospital for Children
Organization: Texas Scottish Rite Hospital for Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU20250837
Record Dates: First submitted 2025-04-25; First posted 2025-05-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: ACL Injuries
Keywords: ACL; menstruation; Neuromuscular training; female athlete
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MC-Synced NTP (Experimental): Menstrual cycle-synced neuromuscular training program
  Interventions: Other: MC-synced NTP
- Blinded NTP (Active Comparator): Blinded neuromuscular training program
  Interventions: Other: Blinded NTP

INTERVENTIONS:
Other: MC-synced NTP — Menstrual cycle-synced neuromuscular training program
  Arms: MC-Synced NTP
Other: Blinded NTP — Blinded neuromuscular training program
  Arms: Blinded NTP

SUMMARY:
This is a research study of female athletes participating in at least one running/cutting sport, who have no current conditions that would limit ability to perform sport-like movement tasks (such as running or jumping), and have reported to be post-menarche (a regular period).

The purpose of this study is to leverage the menstrual cycle (MC) to improve the success of a neuromuscular training program (NTP) that has been shown to reduce high-risk movement patterns in adolescent females. The findings of this study may not only help develop more effective, personalized injury prevention strategies for female athletes, but may also have the potential to reduce ACL injury rates while improving long-term physical activity and health for active females.

The researchers hope that this information may help reduce ACL injury rates and enhance long-term musculoskeletal health in female athletes, while promoting greater equity in sports medicine and performance training.

Participants will be asked to wear an Oura Ring (a ring that is placed on a finger of the non-dominant hand) that will be used to track their menstrual cycle phases. The Oura Ring will be connected using a software called "Natural Cycles", which will sync to either a smart phone via Bluetooth, or data from the device can be downloaded to an iPad utilized by the research team. Participants will also take part in an 8-week Neuromuscular Training Program (NTP), that consists of two 30-minute training sessions per week, which will include dynamic exercises designed to improve strength and power, balance, and stability, as well as help to build a foundation of muscular endurance. Before starting the training program, participants will be asked to complete several questionnaires focused on activity level, sport participation characteristics, sport-related injury history, and menstrual cycle history, and both before and after completing the training program, participant movement patterns may be evaluated. For the training program, participants will be randomized into one of two groups - one that syncs the training type to the participant's menstrual cycle and one that does not. All participants will receive the same exercises, however, a participant's assigned group will determine when they receive certain exercises.

Participation in this study is completely voluntary. Participation is expected to last up to 7 months.

This is a minimal risk research study. There is a small risk of falling during movement tasks, skin irritation from tape that is used during movement evaluation, psychological stress from survey questions, and loss of confidentiality. To minimize these risks, participants may request rest breaks or stop participating at any time. Participants may also refuse to answer any questions that are asked, and all information collected from this research will be stored in a secure electronic database. This information known as "data" will not be shared with any person outside of the study team.

There is no benefit to participants who participate in this research study. However, the investigators hope the information gathered from this research may benefit others in the future.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, female high school athlete who participate in running/pivoting sports (e.g., soccer and basketball)
* Aged 13-19 years
* Participants must also have a mobile phone, personally or via a parent, capable of downloading the Oura Ring app and of syncing to a wearable device via Bluetooth.
* Participants will not be excluded from participation if they report irregular periods (not a typical 28-day cycle) or use of hormonal birth control.

Exclusion Criteria:

Participants will be excluded from enrollment if they:

* Have been diagnosed with any musculoskeletal or neuromuscular condition that would impact their movement patterns or training performance
* Report not yet starting their menses or not currently menstruating (no period in the prior 3 months).
* Females in the general student body who are not an active participant of the school's soccer or basketball program will be excluded from the study.
* Participants will be withdrawn if they become pregnant during the course of the study.

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 148 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Attendance Rate | From beginning to end of 8-week training program
  Rate of attendance at training program
Engagement Rate | From beginning to end of 8-week training program
  Level of engagement throughout participation in training program as rated by the study team on a scale of "Very Dissatisfied" to "Very Satisfied".
Participant feedback survey | From beginning to end of 8-week training program
  Participant feedback on training program through a 3-question participant questionnaire.
Biomechanical risk factors associated with ACL injury during dynamic, sport-related tasks | From beginning to end of 8-week training program
  Changes in biomechanical risk factors associated with ACL injury during dynamic, sport-related tasks as evaluated through changes in motion capture analysis of six dynamic, sport-like tasks (step down tap, drop vertical jump, single leg hop, lateral shuffle, deceleration / plant, run-cut / change-of-direction).

CONTACTS AND LOCATIONS:
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No